CLINICAL TRIAL: NCT00171340
Title: An Open-Label, Randomized, MultiCenter Study to Evaluate the Use of Zolendronic Acid in the Prevention of Cancer Treatment-Related Bone Loss in Postmenopausal Women With Estrogen Positive and/or Progesterone Positive Breast Cancer Receiving Letrozole as Adjuvant Therapy
Brief Title: Zoledronic Acid in the Prevention of Cancer Treatment Related Bone Loss in Postmenopausal Women Receiving Letrozole for Breast Cancer.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CFEM345D2405
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Results first posted 2011-05-26 (Estimated); Last update posted 2012-04-16 (Estimated); Status verified 2012-04

CONDITIONS: Bone Loss; Breast Cancer
Keywords: Bone Loss; Osteopenia; Breast cancer; letrozole; zoledronic acid; postmenopausal
MeSH Terms: conditions — Bone Diseases, Metabolic; Breast Neoplasms | interventions — Zoledronic Acid; Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Upfront Zoledronic Acid (Experimental): Zolendronic acid 4 mg Intravenous (IV) 15 minute infusion every 6 months for 5 years beginning on Day 1. All participants took Letrozole tablets 2.5 mg/day for 5 years beginning on Day 1.
  Interventions: Drug: Zoledronic acid; Drug: Letrozole
- Delayed Zoledronic Acid (Experimental): Zolendronic acid 4 mg Intravenous (IV) 15 minute infusion every 6 months beginning when one of the following occurred: BMD T-score <= -2.0 SD at either the lumbar spine or total hip, any clinical fracture unrelated to trauma or an asymptomatic fracture discovered at the Month 36 visit. All participants took Letrozole tablets 2.5 mg/day for 5 years beginning on Day 1.
  Interventions: Drug: Zoledronic acid; Drug: Letrozole

INTERVENTIONS:
Drug: Zoledronic acid — Zolendronic acid 4 mg Intravenous (IV) 15 minute infusion every 6 months.
  Other Names: ZOL446; Zometa®
Drug: Letrozole — Letrozole tablets 2.5 mg/day taken orally for 5 years.
  Other Names: Femara®

SUMMARY:
Post-menopausal breast cancer patients will receive letrozole 2.5 mg daily for the treatment of breast cancer and will be randomized to a treatment group to receive either upfront zoledronic acid 4 mg IV 15-minute infusion every 6 months or delayed start zoledronic acid 4 mg IV 15-minute infusion every 6 months. Delayed start zoledronic acid will be initiated when either the Bone Mineral Density T-score is below -2 Standard Deviations at either the lumbar spine or hip or any clinical fracture unrelated to trauma or an asymptomatic fracture discovered at the month 36 scheduled visit. Letrozole 2.5 mg will be given daily for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Stage I-IIIa breast cancer
* Postmenopausal or recently postmenopausal
* Recent surgery for breast cancer
* Estrogen Receptor positive and/or progesterone receptor positive hormone receptor status
* No prior treatment with letrozole

Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Metastatic disease
* Invasive bilateral disease
* Clinical or radiological evidence of existing fracture in spine or hip
* Prior treatment with IV bisphosphonates in the past 12 months
* Current treatment with oral bisphosphonates ( must be discontinued within 3 weeks of baseline evaluation)
* Use of Tibolone within 6 months
* Prior use of parathyroid hormone for more than 1 week
* Previous or concomitant malignancy
* Abnormal renal function
* History of disease effecting bone metabolism

Other protocol-defined exclusion criteria may apply.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1065 (Actual)
Dates: Start 2003-05; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (100):
- Argentina (2):
  - Novartis Investigative Site, Buenos Aires
  - Novartis Investigative Site, Rosario Santa Fe
- Australia (4):
  - Novartis Investigative Site, New South Wales
  - Novartis Investigative Site, Perth
  - Novartis Investigative Site, South Australia
  - Novartis Investigative Site, Victoria
- Belgium (5):
  - Novartis Investigative Site, Bonheiden
  - Novartis Investigative Site, Brasschaat
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Leuven
  - Novartis Investigative Site, Wilrijk
- Brazil (2):
  - Novartis Investigative Site, Porto Alegre
  - Novartis Investigative Site, São Paulo
- Novartis Investigative Site, Santiago, Chile
- China (2):
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Shanghai
- Novartis Investigative Site, Medellín, Colombia
- Novartis Investigative Site, Nemocnice, Czechia
- Novartis Investigative Site, Cairo, Egypt
- Finland (2):
  - Novartis Investigative Site, Pori
  - Novartis Investigative Site, Turku
- France (5):
  - Novartis Investigative Site, Bordeaux
  - Novartis Investigative Site, Le Havre
  - Novartis Investigative Site, Montpellier
  - Novartis Investigative Site, Poitiers
  - Novartis Investigative Site, Saint-Cloud
- Germany (18):
  - Novartis Investigative Site, Augsberg
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Ebersberg
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Halberstadt
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Hoyerswerda
  - Novartis Investigative Site, Kassel
  - Novartis Investigative Site, Kiel
  - Novartis Investigative Site, Munich
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Neunkirchen
  - Novartis Investigative Site, Rostock
  - Novartis Investigative Site, Stadthagen
  - Novartis Investigative Site, Stendal
  - Novartis Investigative Site, Trier
  - Novartis Investigative Site, Tübingen
  - Novartis Investigative Site, Wiesbaden
- Novartis Investigative Site, Guatemala City, Guatemala
- Novartis Investigative Site, Hong Kong, Hong Kong
- Italy (12):
  - Novartis Investigative Site, Ancona
  - Novartis Investigative Site, Aviano
  - Novartis Investigative Site, Bergamo
  - Novartis Investigative Site, Catanzaro
  - Novartis Investigative Site, Florence
  - Novartis Investigative Site, Genova
  - Novartis Investigative Site, Meldola
  - Novartis Investigative Site, Modena
  - Novartis Investigative Site, Orbassano Torino
  - Novartis Investigative Site, Perugia
  - Novartis Investigative Site, Torino
  - Novartis Investigative Site, Varese
- Novartis Investigative Site, Distrito Federal, Mexico
- Netherlands (9):
  - Novartis Investigative Site, Almere Stad
  - Novartis Investigative Site, Arnhem
  - Novartis Investigative Site, Ede
  - Novartis Investigative Site, Eindhoven
  - Novartis Investigative Site, Hoogeveen
  - Novartis Investigative Site, Leiden
  - Novartis Investigative Site, Nijmegen
  - Novartis Investigative Site, The Hague
  - Novartis Investigative Site, Utrecht
- New Zealand (2):
  - Novartis Investigative Site, Hamilton
  - Novartis Investigative Site, Wellington
- Peru (3):
  - Novartis Investigative Site, Jesus Maria
  - Novartis Investigative Site, La Victoria
  - Novartis Investigative Site, Surquillo
- Philippines (2):
  - Novartis Investigative Site, Cebu City
  - Novartis Investigative Site, Quezon City
- Novartis Investigative Site, Coimbra, Portugal
- South Korea (2):
  - Novartis Investigative Site, Gyeonggi-do
  - Novartis Investigative Site, Seoul
- Spain (6):
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Córdoba
  - Novartis Investigative Site, Gea de Albarracín
  - Novartis Investigative Site, Ibáñez
  - Novartis Investigative Site, la Masó
  - Novartis Investigative Site, Villaroel
- Switzerland (3):
  - Novartis Investigative Site, Bern
  - Novartis Investigative Site, Locarno
  - Novartis Investigative Site, Lugano
- Taiwan (2):
  - Novartis Investigative Site, Chang-hua
  - Novartis Investigative Site, Taipei
- Thailand (2):
  - Novartis Investigative Site, Bangkok
  - Ratchathew, Khonkaen
- United Kingdom (8):
  - Novartis Investigative Site, Birmingham
  - Novartis Investigative Site, Essex
  - Novartis Investigative Site, Manchester
  - Novartis Investigative Site, New Castle Upon Tyne
  - Novartis Investigative Site, Nottingham
  - Novartis Investigative Site, Plymouth
  - Novartis Investigative Site, Sheffield
  - Novartis Investigative Site, Swansea
- Novartis Investigative Site, Caracas, Venezuela

REFERENCES:
- [Derived] Adams A, Jakob T, Huth A, Monsef I, Ernst M, Kopp M, Caro-Valenzuela J, Wockel A, Skoetz N. Bone-modifying agents for reducing bone loss in women with early and locally advanced breast cancer: a network meta-analysis. Cochrane Database Syst Rev. 2024 Jul 9;7(7):CD013451. doi: 10.1002/14651858.CD013451.pub2. PMID 38979716
- [Derived] Coleman R, de Boer R, Eidtmann H, Llombart A, Davidson N, Neven P, von Minckwitz G, Sleeboom HP, Forbes J, Barrios C, Frassoldati A, Campbell I, Paija O, Martin N, Modi A, Bundred N. Zoledronic acid (zoledronate) for postmenopausal women with early breast cancer receiving adjuvant letrozole (ZO-FAST study): final 60-month results. Ann Oncol. 2013 Feb;24(2):398-405. doi: 10.1093/annonc/mds277. Epub 2012 Oct 9. PMID 23047045

RESULTS

PARTICIPANT FLOW:
Groups:
- Zoledronic Acid 4 mg Upfront: Zolendronic acid 4 mg Intravenous (IV) 15 minute infusion every 6 months for 5 years beginning on Day 1. All participants took Letrozole tablets 2.5 mg/day for 5 years beginning on Day 1.
- Zoledronic Acid 4 mg Delayed: Zolendronic acid 4 mg Intravenous (IV) 15 minute infusion every 6 months beginning when one of the following occurred: BMD T-score <= -2.0 SD at either the lumbar spine or total hip, any clinical fracture unrelated to trauma or an asymptomatic fracture discovered at the Month 36 visit. All participants took Letrozole tablets 2.5 mg/day for 5 years beginning on Day 1.
Period: Overall Study
Arm/Group | Zoledronic Acid 4 mg Upfront | Zoledronic Acid 4 mg Delayed
Started | 532 | 533
Completed | 408 | 398
Not Completed | 124 | 135
Not completed — Adverse Event | 46 | 42
Not completed — Lack of Efficacy | 29 | 41
Not completed — Protocol Violation | 7 | 8
Not completed — Withdrawal by Subject | 22 | 19
Not completed — Lost to Follow-up | 0 | 5
Not completed — Abnormal Laboratory Results | 2 | 0
Not completed — Abnormal Test Procedure Results | 6 | 11
Not completed — No Longer Required Study Drug | 1 | 1
Not completed — Administrative Problems | 5 | 2
Not completed — Death | 6 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Zoledronic Acid 4 mg Upfront | Zoledronic Acid 4 mg Delayed | Total
Number analyzed (Participants) | 532 | 533 | 1065
Age Continuous [Median (Full Range); unit: Years] | 57 ((36-87)) [36 to 87] | 58 ((37-81)) [37 to 81] | 57 [36 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 532 | 533 | 1065
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change in Bone Mineral Density (BMD) of the Lumbar Spine (L2-L4) at 12 Months of Therapy.
Description: Bone Mineral Density (g/cm^2) of the Lumbar Spine (L2-L4) as measured by energy x-ray absorptiometry (DXA).
Time Frame: Baseline, 12 months
Population: The Safety Population consists of all Randomized Patients who received at least 1 dose of study medication.
Measure: Mean (Standard Deviation); unit: Percentage change in BMD
Arm/Group | Zoledronic Acid 4 mg Upfront | Zoledronic Acid 4 mg Delayed
Number analyzed (Participants) | 423 | 418
Percentage change in BMD | 2.208 (3.4194) | -3.617 (4.2151)

2. Secondary Outcome: Percentage Change in Bone Mineral Density (BMD) of the Lumbar Spine (L2-L4) at 2, 3, 4 and 5 Years of Therapy.
Description: Bone Mineral Density (g/cm^2) of the Lumbar Spine (L2-L4) as measured by dual energy x-ray absorptiometry (DXA)
Time Frame: Baseline, 2 years. Baseline, 3 years. Baseline, 4 years. Baseline, 5 years.
Population: The Safety Population consists of all Randomized Patients who received at least 1 dose of study medication. n in each of the categories is the number of participants who had safety data at baseline and the given time point.
Measure: Mean (Standard Deviation); unit: Percentage change in BMD
Arm/Group | Zolendronic Acid 4 mg Upfront | Zolendronic Acid 4 mg Delayed
Number analyzed (Participants) | 525 | 535
Percentage change in BMD
  At 2 years (n=339,343) | 3.463 (4.2691) | -4.601 (5.5273)
  At 3 years (n=313,311) | 3.730 (4.884) | -4.871 (6.271)
  At 4 years (n=290,294) | 3.782 (5.7300) | -5.154 (7.1079)
  At 5 years (n=264,264) | 4.308 (6.0242) | -5.414 (7.6185)

3. Secondary Outcome: Percentage Change in Bone Mineral Density (BMD)of the Lumbar Spine (L1-L4) Over 5 Years of Therapy.
Description: Bone Mineral Density (g/cm^2) of the Lumbar Spine (L1-L4)as measured by dual energy x-ray absorptiometry (DXA)
Time Frame: Baseline, 5 years.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percentage change in BMD
Arm/Group | Zolendronic Acid 4 mg Upfront | Zolendronic Acid 4 mg Delayed
Number analyzed (Participants) | 525 | 535
Percentage change in BMD
  At 12 months (n=360,369) | 2.128 (3.2106) | -3603 (4.1808)
  At 2 years (n=339,343) | 3.300 (4.0700) | -4.521 (5.2624)
  At 3 years (n=313,311) | 3.521 (4.5936) | -4.869 (6.0310)
  At 4 years (n=290,294) | 3.529 (5.5410) | -5.148 (6.8803)
  At 5 years (n=264,264) | 3.898 (5.7995) | -5.427 (7.4818)

4. Secondary Outcome: Percentage Change in Bone Mineral Density (BMD) of the Total Hip at 12 Months, 2 Years, 3 Years, 4 Years and 5 Years After Therapy.
Description: Bone Mineral Density (g/cm^2) of the Lumbar Spine (L2-L4) as measured by dual energy x-ray absorptiometry (DXA)
Time Frame: Baseline, 12 months. Baseline, 2 years. Baseline, 3 years. Baseline, 4 years. Baseline, 5 years.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percentage change in BMD
Arm/Group | Zolendronic Acid 4 mg Upfront | Zolendronic Acid 4 mg Delayed
Number analyzed (Participants) | 525 | 535
Percentage change in BMD
  At 12 months (n=419,434) | 1.222 (2.3257) | -2.239 (3.3614)
  At 2 years (n=394,393) | 1.649 (2.7333) | -2.990 (4.4318)
  At 3 years (n=376,365) | 1.754 (3.1375) | -3.302 (4.8942)
  At 4 years (n=336,349) | 1.716 (3.5228) | -3.922 (5.6505)
  At 5 years (n=306,314) | 1.615 (3.7490) | -4.162 (6.0270)

5. Secondary Outcome: Percentage of Participants With Clinical Fractures at 3 Years of Therapy Which Were Not Present at Baseline
Description: At 3 years of therapy the percentage of participants with fractures as detected by X-ray and/ or bone scan.
Time Frame: Baseline,3 years
Population: The Safety Population consists of all Randomized Patients who received at least 1 dose of study medication.
Measure: Number; unit: Percentage of Participants
Arm/Group | Zoledronic Acid 4 mg Upfront | Zoledronic Acid 4 mg Delayed
Number analyzed (Participants) | 525 | 535
Percentage of Participants | 0.6 | 1.5

ADVERSE EVENTS:
Description: Safety Population = Randomized participants who had received at least one dose of randomized treatment medication.
Groups:
- Zoledronic Acid 4mg Upfront: Zolendronic acid 4 mg Intravenous (IV) 15 minute infusion every 6 months for 5 years beginning on Day 1 and Letrozole tablets 2.5 mg/day for 5 years beginning on Day 1.
- Zolendronic Acid 4mg Delayed: Zolendronic acid 4 mg Intravenous (IV) 15 minute infusion every 6 months beginning when one of the following occurred: BMD T-score <= -2.0 SD at either the lumbar spine or total hip, any clinical fracture unrelated to trauma or an asymptomatic fracture discovered at the Month 36 visit. All participants took Letrozole tablets 2.5 mg/day for 5 years beginning on Day 1.
Arm/Group | Zoledronic Acid 4mg Upfront | Zolendronic Acid 4mg Delayed
Serious Adverse Events (participants affected / at risk) | 133/525 | 124/535
Other Adverse Events (participants affected / at risk) | 477/525 | 486/535
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Zoledronic Acid 4mg Upfront (N=525) | Zolendronic Acid 4mg Delayed (N=535)
Anaemia (Blood and lymphatic system disorders) | 1 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 2 | 0
Angina pectoris (Cardiac disorders) | 3 | 2
Angina unstable (Cardiac disorders) | 1 | 0
Aortic valve incompetence (Cardiac disorders) | 1 | 1
Arrhythmia (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 4
Atrioventricular block complete (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 2
Cardiac failure (Cardiac disorders) | 3 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Cardiomegaly (Cardiac disorders) | 0 | 1
Coronary artery stenosis (Cardiac disorders) | 1 | 0
Cytotoxic cardiomyopathy (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 3 | 1
Myocardial ischaemia (Cardiac disorders) | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 1
Tachyarrhythmia (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 2
Goitre (Endocrine disorders) | 0 | 3
Hyperparathyroidism (Endocrine disorders) | 1 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 1
Cataract (Eye disorders) | 1 | 0
Conjunctival haemorrhage (Eye disorders) | 1 | 0
Diplopia (Eye disorders) | 1 | 0
Eye pain (Eye disorders) | 1 | 0
Glaucoma (Eye disorders) | 1 | 1
Iridocyclitis (Eye disorders) | 2 | 0
Iris cyst (Eye disorders) | 1 | 0
Macular degeneration (Eye disorders) | 1 | 0
Retinal disorder (Eye disorders) | 0 | 1
Vision blurred (Eye disorders) | 1 | 0
Visual acuity reduced (Eye disorders) | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 2
Abdominal strangulated hernia (Gastrointestinal disorders) | 1 | 1
Alcoholic pancreatitis (Gastrointestinal disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 2 | 2
Colitis (Gastrointestinal disorders) | 0 | 1
Colitis ischaemic (Gastrointestinal disorders) | 1 | 0
Colitis ulcerative (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Dental caries (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 2
Diverticulum intestinal (Gastrointestinal disorders) | 0 | 1
Femoral hernia (Gastrointestinal disorders) | 1 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 2
Haemorrhoids (Gastrointestinal disorders) | 1 | 1
Hernial eventration (Gastrointestinal disorders) | 0 | 1
Hiatus hernia (Gastrointestinal disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Intestinal prolapse (Gastrointestinal disorders) | 1 | 0
Melaena (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Peptic ulcer (Gastrointestinal disorders) | 0 | 1
Peritonitis (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 2
Reflux oesophagitis (Gastrointestinal disorders) | 1 | 0
Small intestinal stenosis (Gastrointestinal disorders) | 0 | 1
Splenic artery aneurysm (Gastrointestinal disorders) | 1 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 | 1
Umbilical hernia, obstructive (Gastrointestinal disorders) | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Varices oesophageal (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1
Asthenia (General disorders) | 1 | 0
Chest discomfort (General disorders) | 0 | 1
Chest pain (General disorders) | 2 | 4
Death (General disorders) | 1 | 2
General physical health deterioration (General disorders) | 1 | 0
Impaired healing (General disorders) | 3 | 0
Inflammation (General disorders) | 0 | 1
Pain (General disorders) | 1 | 1
Pyrexia (General disorders) | 5 | 3
Sudden death (General disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 1 | 2
Cholecystitis chronic (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 4 | 10
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 1
Liver disorder (Hepatobiliary disorders) | 1 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 1
Actinomycosis (Infections and infestations) | 1 | 0
Biliary tract infection bacterial (Infections and infestations) | 0 | 1
Breast infection (Infections and infestations) | 1 | 0
Bronchopneumonia (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 2 | 2
Device related infection (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 1
Erysipelas (Infections and infestations) | 2 | 1
Escherichia sepsis (Infections and infestations) | 1 | 1
Gallbladder empyema (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Hepatic infection bacterial (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 1
Incision site cellulitis (Infections and infestations) | 0 | 1
Intervertebral discitis (Infections and infestations) | 0 | 1
Localised infection (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 2
Mastitis bacterial (Infections and infestations) | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 4
Post procedural infection (Infections and infestations) | 0 | 1
Postoperative wound infection (Infections and infestations) | 0 | 1
Pyelonephritis acute (Infections and infestations) | 0 | 1
Respiratory moniliasis (Infections and infestations) | 0 | 1
Scrub typhus (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 1
Sinusitis (Infections and infestations) | 1 | 0
Staphylococcal sepsis (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 4 | 1
Urosepsis (Infections and infestations) | 1 | 1
Wound infection (Infections and infestations) | 1 | 1
Wound infection bacterial (Infections and infestations) | 1 | 0
Accident (Injury, poisoning and procedural complications) | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 2
Back injury (Injury, poisoning and procedural complications) | 0 | 1
Cartilage injury (Injury, poisoning and procedural complications) | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 1
Dislocation of joint prosthesis (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 7 | 7
Femur fracture (Injury, poisoning and procedural complications) | 2 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 1 | 1
Hand fracture (Injury, poisoning and procedural complications) | 2 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 1
Incisional hernia (Injury, poisoning and procedural complications) | 1 | 0
Intentional overdose (Injury, poisoning and procedural complications) | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 2 | 0
Joint sprain (Injury, poisoning and procedural complications) | 1 | 0
Meniscus lesion (Injury, poisoning and procedural complications) | 1 | 0
Muscle rupture (Injury, poisoning and procedural complications) | 0 | 1
Post procedural complication (Injury, poisoning and procedural complications) | 1 | 0
Post procedural fistula (Injury, poisoning and procedural complications) | 1 | 0
Procedural nausea (Injury, poisoning and procedural complications) | 1 | 0
Procedural site reaction (Injury, poisoning and procedural complications) | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 2 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 1
Skin laceration (Injury, poisoning and procedural complications) | 1 | 2
Skull fracture (Injury, poisoning and procedural complications) | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0
Traumatic fracture (Injury, poisoning and procedural complications) | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 2 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 3 | 1
Bone density decreased (Investigations) | 1 | 0
Weight decreased (Investigations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 2
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 1
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Bunion (Musculoskeletal and connective tissue disorders) | 1 | 1
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 | 2
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 3
Ligament disorder (Musculoskeletal and connective tissue disorders) | 1 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Monarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 5 | 7
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 4 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 2
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 2 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 | 1
Tenosynovitis stenosans (Musculoskeletal and connective tissue disorders) | 1 | 0
Trigger finger (Musculoskeletal and connective tissue disorders) | 3 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Benign gastrointestinal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Benign pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Fibroadenoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung adenocarcinoma stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Meningioma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to pleura (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Myeloproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Salivary gland adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Brain stem haemorrhage (Nervous system disorders) | 1 | 0
Carotid artery stenosis (Nervous system disorders) | 0 | 1
Carpal tunnel syndrome (Nervous system disorders) | 2 | 2
Cerebrovascular accident (Nervous system disorders) | 0 | 3
Depressed level of consciousness (Nervous system disorders) | 0 | 1
Facial paresis (Nervous system disorders) | 1 | 0
Haemorrhagic cerebral infarction (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 2 | 1
Hemiparesis (Nervous system disorders) | 1 | 0
Intracranial aneurysm (Nervous system disorders) | 1 | 0
Loss of consciousness (Nervous system disorders) | 0 | 1
Meningorrhagia (Nervous system disorders) | 0 | 1
Migraine (Nervous system disorders) | 1 | 0
Multiple sclerosis relapse (Nervous system disorders) | 1 | 0
Normal pressure hydrocephalus (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 1
Sciatica (Nervous system disorders) | 2 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Agitation (Psychiatric disorders) | 1 | 0
Alcoholic psychosis (Psychiatric disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 2 | 0
Depression (Psychiatric disorders) | 2 | 0
Depression suicidal (Psychiatric disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 1
Mental disorder (Psychiatric disorders) | 0 | 1
Panic attack (Psychiatric disorders) | 1 | 0
Suicide attempt (Psychiatric disorders) | 0 | 1
Calculus ureteric (Renal and urinary disorders) | 2 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 2
Nephrotic syndrome (Renal and urinary disorders) | 1 | 0
Obstructive uropathy (Renal and urinary disorders) | 0 | 1
Renal colic (Renal and urinary disorders) | 0 | 2
Renal failure acute (Renal and urinary disorders) | 0 | 2
Renal impairment (Renal and urinary disorders) | 0 | 1
Stress urinary incontinence (Renal and urinary disorders) | 0 | 1
Breast atrophy (Reproductive system and breast disorders) | 0 | 1
Breast calcifications (Reproductive system and breast disorders) | 0 | 1
Breast fibrosis (Reproductive system and breast disorders) | 0 | 2
Ovarian cyst (Reproductive system and breast disorders) | 1 | 1
Perineal fistula (Reproductive system and breast disorders) | 0 | 1
Rectocele (Reproductive system and breast disorders) | 1 | 0
Uterine enlargement (Reproductive system and breast disorders) | 0 | 1
Uterine polyp (Reproductive system and breast disorders) | 1 | 0
Uterine prolapse (Reproductive system and breast disorders) | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0
Vaginal prolapse (Reproductive system and breast disorders) | 2 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Increased viscosity of bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary vascular disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Skin fibrosis (Skin and subcutaneous tissue disorders) | 0 | 1
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 0 | 1
Physical assault (Social circumstances) | 1 | 0
Femoral arterial stenosis (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 0 | 1
Hypertensive crisis (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 0 | 1
Lymphoedema (Vascular disorders) | 1 | 0
Varicose vein (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Zoledronic Acid 4mg Upfront (N=525) | Zolendronic Acid 4mg Delayed (N=535)
Abdominal pain upper (Gastrointestinal disorders) | 18 | 29
Constipation (Gastrointestinal disorders) | 27 | 31
Diarrhoea (Gastrointestinal disorders) | 24 | 31
Dyspepsia (Gastrointestinal disorders) | 23 | 28
Nausea (Gastrointestinal disorders) | 52 | 55
Asthenia (General disorders) | 36 | 50
Fatigue (General disorders) | 93 | 95
Influenza like illness (General disorders) | 49 | 16
Oedema peripheral (General disorders) | 49 | 47
Pyrexia (General disorders) | 76 | 17
Nasopharyngitis (Infections and infestations) | 35 | 29
Urinary tract infection (Infections and infestations) | 16 | 36
Weight decreased (Investigations) | 31 | 23
Weight increased (Investigations) | 57 | 57
Hypercholesterolaemia (Metabolism and nutrition disorders) | 58 | 60
Arthralgia (Musculoskeletal and connective tissue disorders) | 256 | 251
Back pain (Musculoskeletal and connective tissue disorders) | 78 | 78
Bone pain (Musculoskeletal and connective tissue disorders) | 97 | 64
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 57 | 45
Myalgia (Musculoskeletal and connective tissue disorders) | 68 | 71
Neck pain (Musculoskeletal and connective tissue disorders) | 31 | 19
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 42 | 28
Pain in extremity (Musculoskeletal and connective tissue disorders) | 69 | 80
Dizziness (Nervous system disorders) | 28 | 38
Headache (Nervous system disorders) | 75 | 63
Depression (Psychiatric disorders) | 30 | 44
Insomnia (Psychiatric disorders) | 51 | 38
Cough (Respiratory, thoracic and mediastinal disorders) | 38 | 52
Hot flush (Vascular disorders) | 152 | 163
Hypertension (Vascular disorders) | 55 | 59
Lymphoedema (Vascular disorders) | 41 | 36

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.